CLINICAL TRIAL: NCT01904708
Title: The Effects of an Acute Bout of Moderate Intensity Exercise on Plasma Amino Acids in Subjects With Phenylketonuria
Brief Title: Moderate Intensity Exercise and Phenylketonuria
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Current design not able to measure the outcomes anticipated.
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Melanie B Gillingham, Assistant Professor, Oregon Health and Science University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 9202
Record Dates: First submitted 2013-05-31; First posted 2013-07-22 (Estimated); Last update posted 2014-10-16 (Estimated); Status verified 2014-10

CONDITIONS: Phenylketonuria; PKU
Keywords: Phenylketonuria; PKU; Exercise; Muscle Protein Synthesis; Plasma Phenylalanine concentration
MeSH Terms: conditions — Phenylketonurias; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sedentary Visit (No Intervention): Subjects will do quiet, sedentary activities for 8 hours. Hourly blood draws and breath sampling will be collected. Bolus C13-Lysine will be given at hour 4.
- Exercise Visit (Active Comparator): Subjects will do quiet, sedentary activities until hour 5. Blood and breath samples will be collected. At hour 4, subject will consume a bolus of C13-Lysine and immediately walk on a treadmill at a moderate intensity (exercise at 75% of max heart rate) for 45 minutes.
  Interventions: Other: Acute Moderate Intensity Exercise

INTERVENTIONS:
Other: Acute Moderate Intensity Exercise — Moderate intensity exercise by walking on a treadmill at 75% of max heart rate.
  Arms: Exercise Visit

SUMMARY:
Phenylketonuria (PKU), an inherited genetic disorder, can cause irreversible brain damage, declined executive function, and autistic tendencies unless a phenylalanine (Phe) restricted diet is consistently maintained throughout life. Promoting anabolism, the uptake of free amino acids from the extracellular space, is a key component to maintaining plasma phenylalanine concentrations within treatment range among patients with PKU. Exercise promotes muscle protein synthesis and anabolism, but the effect on blood phenylalanine concentrations in patients with PKU has not been reported.

Our objective is to assess the impact of an acute bout of moderate intensity exercise on protein oxidation and plasma amino acid concentrations, as a potential adjunctive therapy for patients with PKU.

The investigators hypothesize that moderate intensity exercise decreases amino acid oxidation, increases muscle protein synthesis, and promotes tissue uptake of essential amino acids, thereby lowering plasma phenylalanine concentrations in patients with Phenylketonuria.

DETAILED DESCRIPTION:
The indicator amino acid oxidation technique utilizes a carbon labeled isotope (L-[13C]) tracer that is ingested orally and is measured in expired breath. This method is based on the theory that if one essential amino acid is deficient, all other amino acids will be oxidized until a break-point is reached and at that time all amino acids will be incorporated into muscle protein synthesis. Using a randomized crossover design the investigators plan to investigate the effects of an acute bout of moderate intensity treadmill exercise versus sedentary activities on plasma amino acids in four subjects with PKU. The long-term goal of this novel research is to determine if exercise could be used as an adjunctive therapy to improve the management of plasma phenylalanine levels and promote a normal, healthy quality of life among patients with PKU.

Patient Recruitment: Four post-pubertal participants ranging from 14-17 years of age with classical phenylketonuria (PKU), treated at Oregon Health & Science University, will participate in this pilot study. Participants will be recruited during their routine clinic visit at Doernbecher Children's Hospital Metabolic clinic.

Study Design: This randomized crossover clinical trial will compare the effects of moderate intensity exercise and sedentary activities on amino acid oxidation and plasma amino acid pools using the indicator amino acid oxidation technique. Each participant will be studied on two separate occasions over a one-month period.

ELIGIBILITY:
Inclusion Criteria:

* plasma phenylalanine concentration of >1200 micromols at diagnosis
* treated by dietary phenylalanine restriction from early infancy
* willing to participate in this study
* stable BMI of 20-25 for the past 3 months
* currently in average to good physical fitness condition
* physically active 3-4 days per week

Exclusion Criteria:

* previously or are currently taking approved or experimental pharmacologic treatments (i.e.: Biopterin (BH4), sapropterin dihydrochloride (Kuvan), Large Neutral Amino Acids (LNAA), pegylated phenylalanine ammonia lyase (PEG-PAL))
* recent history of weight loss
* endocrine disorder
* pregnant
* anemic
* involved in any other study or research protocol
* participation in a current strength training or performance training regimen

Ages: 14 Years to 17 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2 (Actual)
Dates: Start 2013-05; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Compare plasma phenylalanine concentration of final blood draw during exercise versus sedentary visits. | up to 8 hours
  Compare the final blood sample for phenylalanine concentration from each arm of the study.

SECONDARY OUTCOMES:
Breath Enrichment of C13-Lysine during sedentary and exercise | Hours 1-8 of the study day from each arm.
  Compare the AUC total breath enrichment of C13-Lysine during the sedentary and exercise arms.

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Gillingham, PhD, RD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States